CLINICAL TRIAL: NCT00025493
Title: Single Agent Docetaxel for Metastatic Breast Cancer in Patients Aged 70 Years and Older (and in a Cohort of Patients Younger Than 60 Years)
Brief Title: S0029 Docetaxel in Treating Older Women With Metastatic Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: poor accrual
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068966; U10CA032102 (NIH); S0029 (Other: SWOG)
Record Dates: First submitted 2001-10-11; First posted 2003-01-27 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- docetaxel (Experimental): docetaxel
  Interventions: Drug: docetaxel

INTERVENTIONS:
Drug: docetaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of docetaxel in treating older women who have metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility of treating elderly women with metastatic breast cancer with docetaxel.
* Determine the overall survival, 2-year survival, and response (confirmed and unconfirmed complete and partial) in patients treated with this drug.
* Determine the toxicity and tolerability of this drug in these patients.
* Determine the feasibility of using standardized self-report measures of comorbidity, depression, and functional status in elderly cancer patients.
* Determine the parameters of clinical pharmacology of this drug in elderly patients and in patients under 60 years of age.
* Determine, preliminarily, the genetic polymorphisms and gene expression levels of enzymes involved in drug metabolism and resistance in patients treated with this drug.

OUTLINE: Patients are stratified according to age (70 and over vs under 60).

Patients receive docetaxel IV over 1 hour on day 1. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 3 years.

PROJECTED ACCRUAL: Approximately 80 patients (60 patients age 70 and over and 20 patients under age 60) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed breast cancer

  * Distant metastatic disease confirmed by histology, cytology, or strong clinical evidence
* Measurable disease
* No known brain or CNS metastases
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 70 and over OR
* Under 60

Sex:

* Female

Menopausal status:

* Not specified

Performance status:

* Zubrod 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute granulocyte count at least 1,500/mm^3
* Hemoglobin at least 9 g/dL
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than upper limit of normal (ULN)
* SGOT or SGPT no greater than 1.5 times ULN (2.0 times ULN if liver metastases are present)
* Alkaline phosphatase no greater than 1.5 times ULN (2.0 times ULN if liver metastases are present)

Renal:

* Creatinine no greater than ULN

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* HIV negative
* No other prior malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or adequately treated stage I or II cancer in complete remission

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent immunotherapy for breast cancer

Chemotherapy:

* Prior adjuvant or neoadjuvant chemotherapy allowed
* Prior adjuvant taxanes allowed
* No other concurrent chemotherapy for breast cancer

Endocrine therapy:

* Prior hormonal therapy in the adjuvant setting or for metastatic disease allowed
* No concurrent hormonal therapy for breast cancer

Radiotherapy:

* No concurrent radiotherapy for breast cancer

Surgery:

* Not specified

Other

* No more than 1 prior regimen for advanced, recurrent, or metastatic disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2001-10; Primary Completion 2007-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Study treatment feasibility | monthly for duration of accrual

SECONDARY OUTCOMES:
Overall survival | at weeks 10 and 19, then every 3 months for 3 years
Survival at 2 years | at weeks 10 and 19, then every 3 months for 2 years
Response rate (confirmed and unconfirmed complete and partial response) | at weeks 10 and 19, then every 3 months for 3 years
Toxicity and tolerability | at week 1, then every 3 weeks
Feasibility of standardized self-report measures of comorbidity, depression, and functional status | upon completion of patient accrual
Comparison of clinical pharmacologic parameters between elderly patients and patients under 60 years of age | upon completion of patient accrual

CONTACTS AND LOCATIONS:
Overall Officials: Silvana Martino, DO, Study Chair — Saint John's Cancer Institute